CLINICAL TRIAL: NCT04492176
Title: A Clinical Clinical Observation of CO2 Fractional Laser in Female Vaginal Repair: A Non-randomized, Open, Inter-group and Self-controlled Trial Before and After Treatment
Brief Title: A Clinical Clinical Observation of CO2 Fractional Laser in Female Vaginal Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Gang Wang, MD, chief of dermatology, Xijing Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: XijingH-PF-20190718
Record Dates: First submitted 2019-08-04; First posted 2020-07-30 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Vaginal Atrophy
Keywords: Vaginal atrophy; Vaginal relaxation; stress urinary incontinence; CO2 fractional laser
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CO2 fractional laser（ACUPULSE,Lumenis） (Experimental): gradually withdrawn from inside to outside of vaginal. with CO2 fractional laser therapy ( hexagonal spot , 10-12.5m J/cm2 , density 5-15%，ACUPULSE,Lumenis) ,once a month for a total of 3 times .CO2 fractional laser stimulates fibroblasts to synthesize and secrete collagen fibers, elastic fibers, reticular fibers and organic matrix through dot exfoliation and thermal stimulation, thus thickening the vaginal wall and achieving long-term vaginal tightening effect. The heat effect of CO2 laser can stimulate vasodilation, increase blood flow, increase cell oxidation and nutrients, increase mitochondrial ATP release, activate cell function, enhance vaginal mucosal secretion, enhance secretion, normalize vaginal PH and bacterial flora, and then reduce the probability of gynecological infection.
  Interventions: Device: CO2 fractional laser（ACUPULSE,Lumenis）
- before treatment (No Intervention): the patient did not receive laser treatment

INTERVENTIONS:
Device: CO2 fractional laser（ACUPULSE,Lumenis） — gradually withdrawn from inside to outside of vaginal. with Acupulse Femtouch mode therapy ( hexagonal spot , 10-12.5m J/cm2 , density 5-15%) ,once a month for a total of 3 times
  Arms: CO2 fractional laser（ACUPULSE,Lumenis）

SUMMARY:
1. Vaginal atrophy is the most common indication in the treatment of vaginal rejuvenation. Its main manifestation is vaginal relaxation syndrome, which may be the early symptom of female pelvic floor dysfunction. It is a common gynecological physiological change in women. Its clinical manifestations include vaginal wall relaxation, decreased elasticity, poor dryness sensitivity, internal environment disorder, and so on. Vaginal exhaust, often combined with urinary incontinence, pelvic organ prolapse, chronic pelvic discomfort and other symptoms, seriously affecting patients'health and quality of sexual life. At present, there are many treatments for vaginal relaxation,vaginal constriction and laser therapy are the most effective and widely accepted treatments. Laser therapy with small trauma and short repair time has attracted much attention.
2. CO2 fractional laser (Acupulse) stimulates fibroblasts to synthesize and secrete collagen fibers, elastic fibers, reticular fibers and organic matrix through dot exfoliation and thermal stimulation, thus thickening the vaginal wall and achieving long-term vaginal tightening effect. The heat effect of CO2 laser can stimulate vasodilation, increase blood flow, increase cell oxidation and nutrients, increase mitochondrial ATP release, activate cell function, enhance vaginal mucosal secretion, enhance secretion, normalize vaginal PH and bacterial flora, and then reduce the probability of gynecological infection.
3. It has been reported that CO2 lattice laser can stimulate collagen synthesis and rearrangement. It has also been reported that CO2 lattice laser may have important clinical significance in improving the morphology and function of vaginal epithelial cells.

DETAILED DESCRIPTION:
1. Vaginal atrophy is the most common indication in the treatment of vaginal rejuvenation. Its main manifestation is vaginal relaxation syndrome, which may be the early symptom of female pelvic floor dysfunction. It is a common gynecological physiological change in women. Its clinical manifestations include vaginal wall relaxation, decreased elasticity, poor dryness sensitivity, internal environment disorder, and so on. Vaginal exhaust, often combined with urinary incontinence, pelvic organ prolapse, chronic pelvic discomfort and other symptoms, seriously affecting patients'health and quality of sexual life. At present, there are many treatments for vaginal relaxation,vaginal constriction and laser therapy are the most effective and widely accepted treatments. It should be noted that patients with vaginal constriction need anti-scar training for a long time after operation to prevent the effect of vaginal entrance narrowing and vaginal wall scar formation on the quality of life of patients during the repair period. Therefore, laser therapy with small trauma and short repair time has attracted much attention.
2. CO2 fractional laser (Acupulse) stimulates fibroblasts to synthesize and secrete collagen fibers, elastic fibers, reticular fibers and organic matrix through dot exfoliation and thermal stimulation, thus thickening the vaginal wall and achieving long-term vaginal tightening effect. The heat effect of CO2 laser can stimulate vasodilation, increase blood flow, increase cell oxidation and nutrients, increase mitochondrial ATP release, activate cell function, enhance vaginal mucosal secretion, enhance secretion, normalize vaginal Internal environment and bacterial flora, and then reduce the probability of gynecological infection.
3. It has been reported that CO2 lattice laser can stimulate collagen synthesis and rearrangement. It has also been reported that CO2 lattice laser may have important clinical significance in improving the morphology and function of vaginal epithelial cells. Our center has also passed the clinical observation ethical review of CO2 lattice laser to improve female vaginal relaxation in 2016, and completed the clinical trial at the end of 2017. The data further confirm that CO2 lattice laser can improve vaginal relaxation and is significantly effective for stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Married women aged 25-75 with improvement needs;
* Agree to participate in the experiment and sign the informed consent.
* Female sexual dysfunction patients;
* No other external treatment was performed before treatment at the lesion site.
* VTI instrument was used for intravaginal pressure test to assess urinary incontinence and vaginal senility caused by chronic muscle dysfunction

Exclusion Criteria:

* Pregnant or lactating women;
* suffering from severe mental disorders, psychological disorders, personality disorders and major organ dysfunction;
* Patients with severe hematological diseases, Sjogren's syndrome, systemic and therapeutic site infections;
* Patients who took high doses of anticoagulants or hormones within one month;
* Laser allergy history, photosensitive reactor;
* Women with acute vaginitis or cervicitis;
* Pap smear positive patients;
* Female HIV (HIV), HPV (papillary virus), HSV (herpes simplex virus) positive patients;
* Use of antifungal drugs, vaginal administration, vaginal irrigation and female sprays in the past 30 days
* The condition of the visual field of laser surgery affected by ulceration and infection of the skin lesion
* Those who have undergone vaginal tightening surgery with other substances or means

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
female sexual function FSFI score（Female Sexual Function Index ） | Changes from preoperative to 1 year after initial treatment
  Questionnaire content involving sexual activity, intercourse, sexual stimulation, sexual desire or sexual interest, sexual excitement or sexual arousal, evaluation of female sexual function, questionnaire score ≤ 26.55 is considered female sexual dysfunction
urinary incontinence questionnaire short form assessment | Changes from preoperative to 1 year after initial treatment
  Evaluate urinary incontinence questionnaire short form assessment
VHIS score in vaginal environment | Changes from preoperative to 1 year after initial treatment
  Comprehensive evaluation of vaginal status by vulvar status, internal PH value, vaginal elasticity, guided endocrine secretion, and vaginal moistness
vaginal pressure VTI data detection | Changes from preoperative to 1 year after initial treatment
  Evaluate vaginal pressure by VTI data detection
pelvic floor magnetic resonance MRI plain | Changes from preoperative to 1 year after initial treatment
  Measure tissue structures in the pelvis
scantransvaginal ultrasound | Changes from preoperative to 1 year after initial treatment
  Measure the structures of the vagina
histopathological biopsy | Changes before and 1month after treatment
  5 cases were randomly selected for histopathological biopsy

SECONDARY OUTCOMES:
patient satisfaction assessment | Changes from preoperative to 1 year after initial treatment
  Patient satisfaction: Very satisfied, satisfied, average, dissatisfied, very dissatisfied
VAS Pain Assessment(Immediately after Treatment) | 3 months
  VAS pain scoring criteria (0-10 points): 0 points: no pain; less than 3 points: mild pain, can tolerate; 4 points 1-6 points: patients with pain and affect sleep, can still tolerate; 7 points-10 points : The patient has increasing pain, and the pain is intolerable

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Principal Investigator — Dermatology Derpartment of Xijing Hospital
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China